CLINICAL TRIAL: NCT04686708
Title: Impact of the COVID-19 Pandemic on Emergency General Surgery Outcomes: a Single-center Cohort Study
Brief Title: COVID-19 Pandemic and General Surgery Emergencies
Status: Completed | Type: Observational
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Suleyman Utku Celik, Principal Investigator, Gulhane Training and Research Hospital
Other Study IDs: Gulhane2020-258
Record Dates: First submitted 2020-12-27; First posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Emergencies
Keywords: COVID-19; emergency treatment; general surgery; pandemic
MeSH Terms: conditions — Emergencies; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-pandemic period: Patients managed in the pre-pandemic period
  Interventions: Other: Emergency general surgical admissions
- Pandemic period: Patients managed in the pandemic period
  Interventions: Other: Emergency general surgical admissions

INTERVENTIONS:
Other: Emergency general surgical admissions — All emergency general surgical admissions are admitted initially to the emergency department and then referred to the general surgery department for further management (medical, interventional, or surgical approaches).

SUMMARY:
A retrospective analysis of emergency general surgical admissions during the first six months of the pandemic (from March 11 to September 11, 2020) and the same period in 2019, will be conducted.

DETAILED DESCRIPTION:
The volume and disease severity of emergency general surgery admissions between the first six-month period of the pandemic and the similar time period in the prepandemic period in 2019 will be compared.

Patients admitted during the first six months of the COVID-19 pandemic, from March 11 to September 11, 2020, will be included. As a comparison group, similar data will be collected on patients admitted to the general surgery department during the same period in 2019. Patient and disease characteristics, including demographics, initial leukocyte and C-reactive protein levels, diagnosis, treatment strategies, complications, duration of hospital stay, 30-day rehospitalization rate, and 30-day reoperation rate will be reviewed. Complications will be classified according to Clavien-Dindo classification. Tokyo Guidelines 2018/2013 will be used to assess the severity of the acute cholecystitis.

After the patients are divided into two groups: (1) prepandemic period and (2) pandemic period, descriptive statistics will be presented as the medians and ranges, and frequencies (%). Associations between variables will be evaluated using the Mann-Whitney U test (for continuous variables) or Pearson's chi-square and Fisher exact tests (for categorical variables), where appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Patients admitted during the first six months of the pandemic, from March 11 to September 11, 2020, and patients admitted during the same period in 2019

Exclusion Criteria:

* Patients younger than 18 years
* Patients positive for COVID-19
* Patients required elective surgery
* Patients re-operated because of a postoperative complication of an elective surgical procedure

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consecutive patients admitted during the first six months of the pandemic and patients admitted during the same period in 2019 at the department of general surgery, Gulhane Training and Research Hospital
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-09-11 (Actual)

PRIMARY OUTCOMES:
Incidence of general surgical emergencies | 6 months
  The incidence of surgical emergencies (acute appendicitis, acute cholecystitis, bowel obstruction, incarcerated or strangulated hernia, ulcer perforation, diverticulitis, mesenteric ischemia, acute pancreatitis, abdominal trauma, and perianal abscess) admitted to the general surgery service in the first six months of the pandemic and in the same period in 2019 will be compared separately and together.

SECONDARY OUTCOMES:
Complication rate | 1 month
  30-day complication rates of surgical emergencies will be compared between the prepandemic period and the COVID-19 pandemic period. Complications will be graded according to the Clavien-Dindo classification system.

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Study protocol will be seen on clicaltrials.gov